CLINICAL TRIAL: NCT01096264
Title: Establishment of Local Arterial Stiffness Normal Values (Carotid and Femoral) on Healthy Volunteers Using Supersonic Shear Imaging
Brief Title: Non-Invasive Quantitative Imaging of Human Local Arterial Wall Elasticity Using Supersonic Shear Imaging
Acronym: ULTRAFASTECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: National Research Agency, France (Other); SOCIETE FRANCAISE DE MEDECINE VASCULAIRE (Unknown)
Responsible Party: Dr Emmanuel Messas, Hôpital Européen Georges Pompidou
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 2009-03
Record Dates: First submitted 2010-03-19; First posted 2010-03-31 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers; Vascular Ehlers Danlos Syndrome
Keywords: Arterial stiffness; Pulse wave velocity; Ultrafastecho; Supersonic shear imaging
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteer (Other): Healthy volunteer undergoing two imagery evaluation :
  * SSI technique for local PWV and arterial stiffness evaluation
  * SphygmoCor® for aortic PWV.
  Interventions: Other: SSI and SphygmoCor® evaluations
- vEDS patients (Other): vEDS patients undergoing two imagery evaluations:
  * SSI technique for local PWV and arterial stiffness evaluation
  * SphygmoCor® for aortic PWV.
  Interventions: Other: SSI and SphygmoCor® evaluations

INTERVENTIONS:
Other: SSI and SphygmoCor® evaluations — * SSI evaluation need Aixplorer vascular ultrasound machine (available in our department) with 8 MHz linear array probe applied on the carotid and femoral artery.
  * SphygmoCor® evaluation used pressure captors on carotid and femoral sites to record the intra-arterial pressure wave time delay after QRS wave. After distance calculation between the two sites, Aortic PWV can be derived.

SUMMARY:
Arterial stiffness is associated with increased risk of cardiovascular events and death.

Most of existing technique need dedicated device for arterial stiffness evaluation and indirect calculation of intra arterial pressure. Supersonic Shear Imaging (SSI) is a novel non-invasive technique based on remote palpation of biological tissues that can image with very high temporal resolution (up to 10,000 images/s) and quantify the local viscoelastic properties of tissues. The investigators goal was to apply this SSI technique for arterial stiffness evaluation and local pulse wave velocity (PWV) calculation.

As a first step, the primary goal of this study is to establish normal values of local pulse wave velocity and arterial stiffness (carotid and femoral) by SSI on hundred healthy volunteers.

DETAILED DESCRIPTION:
Provide a more extensive description, if desired. Avoid duplication of information to be recorded elsewhere, such as eligibility criteria or outcome measures.

ELIGIBILITY:
Inclusion criteria for Healthy Volunteers

* Healthy volunteers between 18 and 70 years old of two sexes.
* Caucasian origin
* No tobacco or stopped for more than 5 years
* BMI between 18 and 30 kg/m2.
* Blood pressure after 5 minutes of rest < 140 and 90 mmHg.
* Biological test (haematological biochemistry test in blood , urine test and toxicology tests are all normal) ECG, Blood pressure and Heart rhythm normal.
* All volunteers received information on the research and signed the consent form.
* Health system protection required

Inclusion criteria for patient :

* Age between, 18 et 70 years old for the two sexes
* Presence of two major criteria of Villefranche classification (Am J Med Genet 1998 ;77:31-7) and/or heterozygote pathogen mutation of COL3A1 gene.
* At least 4cm long normal arterial segment (carotid or femoral) analyzed by mode B echograph.
* All patient received information on the research and signed the consent form.
* Health system protection required

General Exclusion Criteria :

* Pregnancy
* Echograph gel allergy
* Local Artery disease (dissection or thrombosis)
* Arrhythmia
* No health insurance coverage
* Incapacity or refused to sign the consent form

Exclusion criteria for Healthy volunteers

* Acute or Chronic Systemic disease (atherosclerosis)
* Alcohol abuse or drug abuse (cocaine,cannabis,etc..)
* Active or past tobacco
* Hypercholesterolemia (LDLc >1.09 g/l)
* Exclusion period according to the national record for volunteer of clinical trial.

Exclusion criteria for Patients

* No intact (carotid or femoral) segment for SSI analysis
* AT2 inhibitors or Beta blockers treatment will be notified but are not considered as exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Normal Values by SSI | day one
  Normal Values by SSI of local PWV and arterial wall stiffness(carotid and femoral).

SECONDARY OUTCOMES:
repeatability of the "primary outcome measure" | Day one
  Evaluation of the repeatability of the "primary outcome measure" on 100 healthy volunteers and 30 patients with Vascular Ehlers Danlos Syndrome (vEDS).
Comparison between 2 populations of values by SSI | Day one
  Comparison between healthy volunteers and vEDS patients for PWV and arterial stiffness evaluated by SSI.
Comparison of values between SSI and standard gold | Day one
  Concordance evaluation between PWV calculated by SSI and Aortic Pulse wave velocity calculated by ShygmoCor®

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Messas, MD, Principal Investigator — Hôpital Européen Georges-Pompidou; Anne Blanchard, MD, Study Chair — Hôpital Européen Georges-Pompidou; Joseph Emmerich, MD, PhD, Study Chair — Hôpital Européen Georges-Pompidou; Xavier Jeunemaitre, MD, PhD, Study Chair — Hôpital Européen Georges-Pompidou; Michael Franck, MD, Study Chair — Hôpital Européen Georges-Pompidou; Olivier Steinchen, MD, Study Chair — Hôpital Européen Georges-Pompidou; Michel Azizi, MD, PhD, Study Chair — Hôpital Européen Georges-Pompidou
Locations (1):
- CIC - Hôpital Européen Georges Pompidou, Paris, France